CLINICAL TRIAL: NCT02062489
Title: Evaluation of Tamoxifen's Efficacy for ER/PR Negative,ER-beta Positive Operable Breast Cancer Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Erwei Song, M.D., Ph.D., Vice President of Sun Yat-Sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCCT2014001
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: breast cancer,; tamoxifen,; ER/PR negative, ER-beta positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tamoxifen (Active Comparator): 20mg(2#)/day, PO, daily, five years
  Interventions: Drug: Tamoxifen
- Placebo (Placebo Comparator): 2#/day, PO, daily, five years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamoxifen — 20 mg(2#)/day, PO, daily
  Other Names: Nolvadex
  Arms: Tamoxifen
Drug: Placebo — 2#/day, PO, daily
  Arms: Placebo

SUMMARY:
The current study is a multicentre, randomized,double-blind, prospective clinical trial stratified patients by the HER2 status of their cancer (negative or positive) which is sponsored by the researchers. The trial is designed to evaluate the effectiveness of tamoxifen as adjuvant therapy for ER(ER-α)/PR negative, ER-β positive operable breast cancer patients. 688 female ER(ER-α)/PR negative, ER-β(wild type ER-β1) positive operable breast cancer patients who had undergone neoadjuvant chemotherapy or directly modified radical mastectomy or breast-conserving surgery were randomly (1:1) enrolled to receive tamoxifen (20 mg per day) or placebo (2# per day) within 6 weeks after postoperative chemotherapy and/or radiation therapy if needed (according to 2013 NCCN breast cancer guideline). If the breast tumor's HER2 is positive, the patient can receive targeted therapy (Herceptin) combined with tamoxifen or placebo. The follow-up time will be eight years. The aim of this trial is to evaluate the effectiveness of tamoxifen as adjuvant therapy for ER(ER-α)/PR negative, ER-β positive operable breast cancer patients by comparing the DFS and OS between tamoxifen group and placebo group and to determine whether the percentage of positive ER-β expression is associated with the response to the hormone therapy in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patients signed the written informed consent
* The patients present with operable unilateral invasive breast cancers without distant metastasis(stage I, II, and III)
* The breast tumor's positive ER/PR rate is <1%, and positive ER-beta1 rate is ≥10% by IHC.
* The patients have no history of neoadjuvant hormone therapy.
* The patients have normal cardiac functions by echocardiography.
* The patients' ECOG scores are ≤0-2.
* Female patient who is ≥ 18yrs, and ≤ 70yrs.
* The patients are non-pregnant, and disposed to practice contraception during the whole trial.
* The patients underwent neoadjuvant chemotherapy plus surgery or directly modified radical mastectomy or breast-conserving surgery (plus sentinel lymph node biopsy or axillary lymph node dissection) after diagnosis of breast cancer.
* The patients underwent chemotherapy, radiation therapy or targeted therapy(herceptin) after surgery according to the 2013 NCCN guideline.
* The results of patients' blood tests are as follows:

Hb≥90g/L; WBC≥4.0×109/L; Plt≥100×109/L; Neutrophils≥1.5×109/L; ALT and AST ≤ triple of normal upper limit; TBIL ≤ 1.5 times of normal upper limit; Creatinine ≤ 1.25 times of normal upper limit.

Exclusion Criteria:

* The patients have other cancers at the same time or have the history of other cancers except controlled skin basal cell carcinoma or skin squamous cell carcinoma or carcinoma in situ of cervix uterus;
* The patients have active infections that were not suitable for chemotherapy;
* The patients have severe non-cancerous diseases.
* The patients have history of neoadjuvant hormone therapy.
* The patients have bilateral breast cancers or DCIS or metastatic breast cancers.
* The patients are undergoing current administration of anti-cancer therapies, or are attending other clinical trials.
* The patients are pregnant or lactational, or they refuse to practice contraception during the whole trial.
* The patients are in some special conditions that they can't understand the written informed consent, such as they are demented or hawkish.
* The patients have allergic history or contraindication of tamoxifen.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival of patients | within 10 years after diagnosis

SECONDARY OUTCOMES:
Rates of adverse reactions | within 5 years when patients is undergoing tamoxifen or placebo treatment
Distant metastasis-free survival | within 10 years after diagnosis
Overall survival | within 10 years after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Erwei Song, M.D.,Ph.D., Study Chair — Sun Yat-Sen Memerial Hospital of Sun Yat-Sen University; Qiang Liu, MD.PhD., Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (17):
- China (17):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Women and Children Hospital, Guangzhou, Guangdong
  - Guangzhou Army General Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangzhou Women and Children Hospital, Guangzhou, Guangdong
  - The third people's Hospital of Huizhou, Huizhou, Guangdong
  - Xinjiang Medical School Cancer Center, Xinjiang, Xinjiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Dongguan People's Hospital, Dongguan
  - Foshan First People's Hospital, Foshan
  - The sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Lian Jiang People's Hospital, Lianjiang
  - The Third Hospital of Nanchang, Nanchang
  - The Second People's Hospital of Shenzhen, Shenzhen